CLINICAL TRIAL: NCT00990834
Title: Muscle Characteristics Associated With Statin Therapy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit subjects.
Sponsor: Scripps Health (Other)
Responsible Party: Truong, H. Tam, MD, Scripps Mercy Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MCAST
Record Dates: First submitted 2009-10-05; First posted 2009-10-07 (Estimated); Last update posted 2015-05-22 (Estimated); Status verified 2015-05

CONDITIONS: Hydroxymethylglutaryl-CoA Reductase Inhibitors; Myopathy
Keywords: Statin; Myopathy; Hydroxymethylglutaryl-CoA Reductase Inhibitors; Atrogin-1
MeSH Terms: conditions — Muscular Diseases | interventions — Simvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Statin exposure (Experimental): Subjects' endpoints will be measured before and after one to eight months of statin exposure.
  Interventions: Drug: simvastatin

INTERVENTIONS:
Drug: simvastatin — simvastatin 80 mg PO daily for one to eight months.
  Other Names: Zocor

SUMMARY:
The purpose of this study is to investigate the mechanism of statin-related myopathy by evaluating muscle samples before and after statin exposure.

DETAILED DESCRIPTION:
Statins have been proven to reduce cardiovascular events and mortality in large clinical trials but remain underutilized partly due to the associated myopathy. Severe reactions manifested as rhabdomyolysis are rare but myalgia is commonly noted in clinical practice. The pathophysiology of these events remains obscure. Previous studies suggest that statins block the downstream products (such as cellular signaling molecules) of the mevalonate pathway needed for normal muscle function. Other studies show that statins are associated with gene expressions involved in muscle damage such as atrogin-1. We will quantify these entities pre and post statin therapy to better understand these reactions.

ELIGIBILITY:
Inclusion Criteria:

* Primary surgeon's permission.
* Patient is > 21 years of age.
* Patient will go through a two phase surgery with the two procedures one to eight months apart.
* Patient or representative understands the nature of the study.
* Normal thyroid stimulating hormone (TSH).
* LDL-cholesterol > 100 mg/dL or highly sensitive C-reactive protein (hsCRP) > 2.0.
* One of the following risk factors: male > 45 year old or female > 55 year old, smoker, hypertension, first degree family history of coronary artery disease < 55 year old, HDL <40 mg/dL, chronic kidney disease, diabetes mellitus, previous TIA or stroke, previous coronary artery disease.

Exclusion Criteria:

* Has been on a lipid-lowering medication previously.
* Severe illness (e.g. trauma or sepsis) more than 24 hours before obtaining the first biopsy.
* Less than a 10% reduction of LDL after 3 months of therapy (indicative of non-adherence).
* Contraindications to statins such as liver failure.
* History of underlying muscle disorder.
* Taking amiodarone.

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-11; Primary Completion 2011-06 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Atrogin-1 expression. | One to eight months.
Intramuscular Ras level. | One to eight months.

SECONDARY OUTCOMES:
Intramuscular Coenzyme Q10 level. | One to eight months.
Intramuscular mitochondrial to nuclear DNA ratio. | One to eight months.
Intramuscular geranylgeranylpyrophosphate. | One to eight months.
PPAR-gamma coactivator-1-alpha expression. | One to eight months.

CONTACTS AND LOCATIONS:
Overall Officials: Tam H Truong, MD, Principal Investigator — Scripps Health; Paul S Phillips, MD, Principal Investigator — Scripps Health
Locations (1):
- Scripps-Mercy Hospital, San Diego, California, United States

REFERENCES:
- [Background] Shepherd J, Cobbe SM, Ford I, Isles CG, Lorimer AR, MacFarlane PW, McKillop JH, Packard CJ. Prevention of coronary heart disease with pravastatin in men with hypercholesterolemia. West of Scotland Coronary Prevention Study Group. N Engl J Med. 1995 Nov 16;333(20):1301-7. doi: 10.1056/NEJM199511163332001. PMID 7566020
- [Background] Long-Term Intervention with Pravastatin in Ischaemic Disease (LIPID) Study Group. Prevention of cardiovascular events and death with pravastatin in patients with coronary heart disease and a broad range of initial cholesterol levels. N Engl J Med. 1998 Nov 5;339(19):1349-57. doi: 10.1056/NEJM199811053391902. PMID 9841303
- [Background] Kashani A, Phillips CO, Foody JM, Wang Y, Mangalmurti S, Ko DT, Krumholz HM. Risks associated with statin therapy: a systematic overview of randomized clinical trials. Circulation. 2006 Dec 19;114(25):2788-97. doi: 10.1161/CIRCULATIONAHA.106.624890. Epub 2006 Dec 11. PMID 17159064
- [Background] Bruckert E, Hayem G, Dejager S, Yau C, Begaud B. Mild to moderate muscular symptoms with high-dosage statin therapy in hyperlipidemic patients--the PRIMO study. Cardiovasc Drugs Ther. 2005 Dec;19(6):403-14. doi: 10.1007/s10557-005-5686-z. PMID 16453090
- [Background] Flint OP, Masters BA, Gregg RE, Durham SK. Inhibition of cholesterol synthesis by squalene synthase inhibitors does not induce myotoxicity in vitro. Toxicol Appl Pharmacol. 1997 Jul;145(1):91-8. doi: 10.1006/taap.1997.8131. PMID 9221828
- [Background] Nishimoto T, Ishikawa E, Anayama H, Hamajyo H, Nagai H, Hirakata M, Tozawa R. Protective effects of a squalene synthase inhibitor, lapaquistat acetate (TAK-475), on statin-induced myotoxicity in guinea pigs. Toxicol Appl Pharmacol. 2007 Aug 15;223(1):39-45. doi: 10.1016/j.taap.2007.05.005. Epub 2007 May 24. PMID 17599378
- [Background] Matzno S, Yasuda S, Juman S, Yamamoto Y, Nagareya-Ishida N, Tazuya-Murayama K, Nakabayashi T, Matsuyama K. Statin-induced apoptosis linked with membrane farnesylated Ras small G protein depletion, rather than geranylated Rho protein. J Pharm Pharmacol. 2005 Nov;57(11):1475-84. doi: 10.1211/jpp.57.11.0014. PMID 16259781
- [Background] Young JM, Florkowski CM, Molyneux SL, McEwan RG, Frampton CM, George PM, Scott RS. Effect of coenzyme Q(10) supplementation on simvastatin-induced myalgia. Am J Cardiol. 2007 Nov 1;100(9):1400-3. doi: 10.1016/j.amjcard.2007.06.030. Epub 2007 Aug 16. PMID 17950797
- [Background] Draeger A, Monastyrskaya K, Mohaupt M, Hoppeler H, Savolainen H, Allemann C, Babiychuk EB. Statin therapy induces ultrastructural damage in skeletal muscle in patients without myalgia. J Pathol. 2006 Sep;210(1):94-102. doi: 10.1002/path.2018. PMID 16799920
- [Background] Grundy SM, Cleeman JI, Merz CN, Brewer HB Jr, Clark LT, Hunninghake DB, Pasternak RC, Smith SC Jr, Stone NJ; National Heart, Lung, and Blood Institute; American College of Cardiology Foundation; American Heart Association. Implications of recent clinical trials for the National Cholesterol Education Program Adult Treatment Panel III guidelines. Circulation. 2004 Jul 13;110(2):227-39. doi: 10.1161/01.CIR.0000133317.49796.0E. PMID 15249516
- [Background] Sever PS, Dahlof B, Poulter NR, Wedel H, Beevers G, Caulfield M, Collins R, Kjeldsen SE, Kristinsson A, McInnes GT, Mehlsen J, Nieminen M, O'Brien E, Ostergren J; ASCOT investigators. Prevention of coronary and stroke events with atorvastatin in hypertensive patients who have average or lower-than-average cholesterol concentrations, in the Anglo-Scandinavian Cardiac Outcomes Trial--Lipid Lowering Arm (ASCOT-LLA): a multicentre randomised controlled trial. Lancet. 2003 Apr 5;361(9364):1149-58. doi: 10.1016/S0140-6736(03)12948-0. PMID 12686036
- [Background] Cohen JC, Boerwinkle E, Mosley TH Jr, Hobbs HH. Sequence variations in PCSK9, low LDL, and protection against coronary heart disease. N Engl J Med. 2006 Mar 23;354(12):1264-72. doi: 10.1056/NEJMoa054013. PMID 16554528
- [Background] Hanai J, Cao P, Tanksale P, Imamura S, Koshimizu E, Zhao J, Kishi S, Yamashita M, Phillips PS, Sukhatme VP, Lecker SH. The muscle-specific ubiquitin ligase atrogin-1/MAFbx mediates statin-induced muscle toxicity. J Clin Invest. 2007 Dec;117(12):3940-51. doi: 10.1172/JCI32741. PMID 17992259
- [Background] Shishehbor MH, Patel T, Bhatt DL. Using statins to treat inflammation in acute coronary syndromes: Are we there yet? Cleve Clin J Med. 2006 Aug;73(8):760-6. doi: 10.3949/ccjm.73.8.760. PMID 16913201